CLINICAL TRIAL: NCT03086694
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital
Brief Title: Goal-Directed Fluid Therapy for Patients Undergoing Oro-Maxillofacial Surgery
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(II)_20160110
Record Dates: First submitted 2017-02-06; First posted 2017-03-22 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2017-03

CONDITIONS: Blood Pressure, Low
Keywords: oromaxillofacial surgery; nasotracheal intubation; stroke volume variation
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group surgery: using medications to maintain low stable blood pressure

SUMMARY:
Orthognathic surgery, one kind of Oro-maxillofacial surgery, is a complicate surgery that undergoes several hours with nasotracheal intubation general anesthesia. To limit blood loss during operation, the patients are often under intentional hypotension. However, the intentional hypotension may confuse with hypovolemic induced low blood pressure. The hypothesis is using flotrac (to measure stroke volume variation) to keep the patients hemodynamics stable under Tridil and propofol infusion and avoid over-infusion of crystalloid or colloid and prevent hypovolemia induced postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Orthognathic surgery, one kind of oro-maxillofacial surgery, is a complicated surgery that undergoes several hours with nasotracheal intubation general anesthesia. Patients without premedication undergo orthognathic surgery with nasotracheal intubation general anesthesia.

Patients without premedications Monitoring of patients with entropy for consciousness, ECG, with noninvasive BP and invasive blood pressure through redial artery, train-of-four monitor, target controlled infusion of propofol, infusion Tridil, and sevoflurane for mainly anesthesia maintenance. Ventilator setting as volume control (8-12ml/kg), frequency respiratory rate (8-12/min), I/E ratio: 1/2, positive end expiratory pressure: 4 mmHg, Fraction inspiratory O2: 60%.

To maintain the MAP >60-55 mmHg, urine output 0.5-1ml/kg, and body core temperature > 36 Celsius degree.

Closely observation of patients postoperatively for adverse events or complications.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo orthognathic surgery, ASA I~III, 20 to 65 years old, no mouth limitation

Exclusion Criteria:

* ankylosing spondylitis, limited mouth opening < 3 cm, liver or renal disease, obese patients (BMI>35kg/m2), patients refused

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who need to operate for abnormal face or abnormal teeth biting
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
blood loss measurement | 10hrs
  to maintain low blood pressure (MAP > 55mmHg) to limit blood loss

SECONDARY OUTCOMES:
assessment of inappropriate fluid infusion | 10hours
  count the fluid given by stroke volume variation but fixed time administration
postoperative adverse events | 2 days
  adequate medications to maintain low stable BP to decrease tissue edematous change

CONTACTS AND LOCATIONS:
Overall Officials: kuang I Cheng, MD, PhD, Principal Investigator — Department of Anesthesiology, Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Department of Anesthesiology, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MC, Tseng KY, Shen YC, Lin CH, Hsu CW, Hsu HJ, Lu IC, Cheng KI. Nasotracheal intubation in patients with limited mouth opening: a comparison between fibreoptic intubation and the Trachway(R). Anaesthesia. 2016 Jan;71(1):31-8. doi: 10.1111/anae.13232. Epub 2015 Oct 12. PMID 26460721